CLINICAL TRIAL: NCT05896098
Title: Effectiveness of Ultrasonography for the Evaluation of Difficult Airway in Obese Patients.
Brief Title: Use of USG in Difficult Airway in Obese
Status: Completed | Type: Observational
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Nazan KOCAOGLU, Assistant Professor, Balikesir University
Other Study IDs: 2020/16
Record Dates: First submitted 2023-05-10; First posted 2023-06-09 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Obesity
Keywords: obesity ultrasound difficult airway
MeSH Terms: conditions — Obesity | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Easy laryngoscopy: Cormack Lehane Classification 1-2a
  Interventions: Other: Ultrasound
- Difficult laryngoscopy: Cormack Lehane Classification 2b-3-4
  Interventions: Other: Ultrasound

INTERVENTIONS:
Other: Ultrasound — Measurement of the airway by ultrasound in obese patients.

SUMMARY:
Introduction and Purpose: Obesity is an increasing public health problem all over the world. Obesity is a proinflammatory multisystemic disease defined as hypertrophy and/or hyperplasia of adipose tissue. Obesity is frequently encountered in elective and emergency surgical procedures and causes more difficulties in airway management. Difficult airway, characterized by difficult mask ventilation and difficult intubation, is especially common in obese and morbidly obese patients. Some studies show that the measurement of anterior neck soft tissue thickness at the level of the vocal cords plays an important role in estimating difficult laryngoscopy in obese patients. Difficult intubation is envisaged in patients with pretracheal soft tissue thickness of 28 mm and neck circumference of more than 50 cm at the level of the vocal cord.

In this prospective observational study, it is aimed to measure the preoperative anterior cervical soft tissue thickness with 3 parameters by USG in obese patients undergoing elective surgery, and to evaluate the relationship of these values with the Han Scale and Cormack-Lehane classification and their effectiveness as an indicator of difficult airway.

DETAILED DESCRIPTION:
Materials and Methods: 157 patients who will undergo elective surgery under general anesthesia, ages between 18-80, BMI ≥ 30 kg/m2, ASA I-II were included in the study. During the preoperative evaluation, patients' gender, age, height, weight, type of surgery, BMI, neck circumference, thyromental distance (TMM), sternomental distance (SMM), hyomental distance (HMM), neck extension, mouth opening and distance between incisors were measured and tooth structure was evaluated. OSAS was evaluated based on the ASA physical condition score and AHI. Mallampati Classification was recorded. Upper lip bite test was performed. Ultrasonographic measurements were made with the patient in the supine position and the head and neck in a neutral position. The Han Scale was used to evaluate difficult mask ventilation. The laryngoscopy image was evaluated and recorded with the Cormack-Lehane Classification, and ≥2b was accepted as difficult laryngoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery, ages between 18-80 BMI over 30, ASA I-II

Exclusion Criteria:

* Facial and cervical trauma, head and neck malignancy, tracheostomy and thyroid surgery, non-cooperate patients, parturients, difficult airway history.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: obese elective surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Difficult laryngoscopy | preoperative evaluation
  To determine the difficult airway in obese patients with 3 levels of anterior soft tissue measurement (cm) with ultrasound.

SECONDARY OUTCOMES:
Difficult mask ventilation | preoperative evaluation
  To determine the difficult airway in obese patients with 3 levels of anterior soft tissue measurement (cm) with ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Nazan Kocaoglu, Principal Investigator — Balikesir University
Locations (2):
- Turkey (Türkiye) (2):
  - Balikesir University, Balıkesir
  - Medical faculty, Balıkesir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ultrasound As A New Tool In The Assessment Of Airway Difficulties: An Observational Study. — https://pubmed.ncbi.nlm.nih.gov/31742568/
- See also: Development of a scoring system for predicting difficult intubation using ultrasonography — https://pubmed.ncbi.nlm.nih.gov/32346164/
- Available data/document: Study Protocol — https://pubmed.ncbi.nlm.nih.gov/14616599/

DOCUMENTS (1):
  • Study Protocol (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/98/NCT05896098/Prot_000.pdf